CLINICAL TRIAL: NCT03431545
Title: An Integrative Approach to Improve Child Outcomes Through Research-based Parent and Teacher Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Susan Landry, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSC-MS-15-0841
Record Dates: First submitted 2018-02-06; First posted 2018-02-13 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Growth & Development
MeSH Terms: interventions — Patj protein, rat

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PALS and BEECH (Experimental): Play and Learning Strategies (PALS) and Beginning Education: Early Childcare at Home (BEECH) include web-based parent and teacher training courses with remote coaching and in-person meetings that support the adults' developing a set of core behaviors that comprise a responsive interactive style including responses contingent to children's needs and interests with rich language input.
  Interventions: Behavioral: PALS and; Behavioral: BEECH
- Control condition (Active Comparator): Parents and teachers conduct business as usual in regards to care-giving in the school and at home.
  Interventions: Behavioral: Control condition

INTERVENTIONS:
Behavioral: PALS and — Play and Learning Strategies (PALS) include web-based parent training courses with remote coaching and in-person meetings that support the adults' developing a set of core behaviors that comprise a responsive interactive style including responses contingent to children's needs and interests with rich language input.
  Parents will begin their 11 week (infant) or 14 week (toddler) parenting program in October and complete it by April. There will be monthly Parent Meetings related to the content they are learning online. Post-assessments will occur in late April and May. Each weekly online parent session will take approximately 30 minutes to complete with a 40 - 60 minute weekly remote coach call.
  Arms: PALS and BEECH
Behavioral: BEECH — Beginning Education: Early Childcare at Home (BEECH) includes web-based teacher training courses with remote coaching and in-person meetings that support the adults' developing a set of core behaviors that comprise a responsive interactive style including responses contingent to children's needs and interests with rich language input.
  Teachers will complete the 20 online sessions weekly, except for planned center closings due to holidays or agency-related events. The three in-person trainings will occur before Session 1 and after Sessions 8 and 14. Each weekly online teacher session will take approximately one-hour for a teacher to complete with a 30 minute weekly remote coach call. Each in-person teacher training will be 6-hours in duration.
  Arms: PALS and BEECH
Behavioral: Control condition — Parents and teachers conduct business as usual in regards to care-giving in the school and at home.
  Arms: Control condition

SUMMARY:
The purpose of this study is to learn whether a combination of two research-proven programs, a responsive caregiving parenting program and a teacher training program, will have an effect on infants' and toddlers' language, cognitive, social-emotional, and self-regulation skills. The interventions are designed to specifically target parent use of a responsive, stimulating caregiving style in the home in combination with teacher instructional practices and the use of a responsive interactive style in the classroom.

ELIGIBILITY:
Inclusion Criteria:

* Given that the target population includes EHS agencies, low-income children speaking English and/or Spanish will be eligible for participation.
* In some cases, children with mild delays (e.g., receiving speech therapy services) can participate.

Exclusion Criteria:

* Children with significant developmental disabilities (e.g., intellectual disabilities, significant sensory impairments, and children diagnosed with moderately severe forms of Autism Spectrum Disorders) will not be consented for assessments as the interventions are not specialized to meet the needs of these children.
* Children primarily speaking a language other than Spanish or English will be excluded due to the fact that appropriate assessment procedures are lacking.
* In terms of exclusionary criteria for teachers, those that are participating in other research studies, or who have recently completed other similar studies, will not be recruited.

Ages: 5 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 260 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2019-09-19 (Actual)

PRIMARY OUTCOMES:
Change in teacher behavior as assessed by the The Quality of Caregiver-Child Interactions for Infant and Toddlers (Q-CCIIT) Scale | baseline, 9 months
  Scales: Support for Social Emotional Development (ratings range from 1 to 7 with higher values indicate better outcome), Support for Language and Literacy (ratings range from 1 to 7 with higher values indicate better outcome), Support for Cognitive Development (ratings range from 1 to 7 with higher values indicate better outcome), Areas of Concern (ratings range from 1 to 3 with higher values indicate worse outcome)
Change in parent behavior as assessed by coding of videotaped parent-child interactions during toy play in the home | baseline, 9 months
  The parent-child dyad will be provided with a set of age-appropriate toys to use during a 15 minute period where parents are asked to play with their children in "typical ways" with a few constraints (e.g., television must be off). Specific variables in each of the four responsiveness components (i.e., support of children's signals and interests, contingent responsiveness, rich language input, warm sensitivity) will be coded from the activity using a previously developed coding system for videotaped parent-child interactions.
Change in parent behavior as assessed by coding of videotaped parent-child interactions during shared reading in the home | baseline, 9 months
  Parent and child will be asked to engage in a 5 minute shared reading activity using books provided to family. Specific variables in each of the four responsiveness components (i.e., support of children's signals and interests, contingent responsiveness, rich language input, warm sensitivity) will be coded from the activity using a previously developed coding system for videotaped parent-child interactions.
Change in child language as assessed by the Preschool Language Scale-Fifth Edition | baseline, 9 months
  Auditory Comprehension Scale (standard scores range from 50 - 150 with higher value representing a better outcome)
Change in child language as assessed by the Early Communication Indicator | baseline, 9 months
Change in child language as assessed by the MacArthur-Bates Communicative Development Inventories - Short Form (parent reported) | baseline, 9 months
Change in child cognitive skills as assessed by the Bayley Scales of Development - III Screening Test | baseline, 9 months
  Cognitive Scale (cut score based on child's chronological age places child in either 'at-risk,' 'emerging,' and 'competent' category)
Change in child social-emotional behaviors as assessed by coding of videotaped parent-child interactions during toy play in the home. | baseline, 9 months
  Children's social behaviors in the home will be coded for: 1) cooperation, 2) language use, 3) social engagement, and 4) initiative during parent-child home-based "free play" interaction.
Change in child social-emotional behaviors as assessed by coding of videotaped parent-child interactions during c in the home. | baseline, 9 months
  Children's social behaviors in the home will be coded for: 1) cooperation, 2) language use, 3) social engagement, and 4) initiative during parent-child home-based "shared reading" interaction.
Change in child socio-emotional skills as assessed by the Brief Infant Toddler Social Emotional Assessment (parent reported) | baseline, 9 months
Change in child self-regulation as assessed by a delay task | baseline, 9 months
  A delay task will be administered to children 24 months and older. In the "Gift/Waiting for the Bow" paradigm the child is left alone for 3 minutes with the gift while the examiner gets a bow (actually, the experimenter will turn his/her back and engage in other activities) and is told not to touch or open the gift; latencies to touching and opening are recorded.
Change in child self-regulation as assessed by a slowing down motor task | baseline, 9 months
  A slowing down motor task will be administered to children 18 months and older. In the "Walk the Line" task, the child walks as slowly as possible down a 6 foot tape line on the floor to their parent; times for a baseline trial (child walk to parent as they normally would) and two slow trials are recorded live. This measure taps early inhibitory control, particularly the ability to modulate a response to context.
Change in child self-regulation as assessed by a suppressing/initiating a response task | baseline, 9 months
  A suppressing/initiating a response task will be administered to children 22 months and older. In the "Tower" task the child and the experimenter build a tower together out of big, foam blocks. The experimenter explains to the child what it means to "take turns." The experimenter then deliberately waits for the child to indicate that the experimenter may have a turn. This task also taps early inhibitory control, particularly the ability to inhibit a desired response (to place the block oneself), in favor of a more socially desirable response (give the experimenter a turn).

SECONDARY OUTCOMES:
Change in teacher characteristics as assessed by the Center for Epidemiologic Studies Depression Scale - Revised | baseline, 9 months
  One depression scale (range from 0 - 4 with higher values related to worse outcomes)
Change in teacher characteristics as assessed by the Parental Modernity Scale | baseline, 9 months
  Two subscales: traditional beliefs (ratings from 1 - 5 with higher values representing traditional beliefs) and progressive beliefs (ratings from 1 - 5 with higher values representing progressive beliefs).
Change in parent characteristics as assessed by the Center for Epidemiologic Studies Depression Scale - Revised | baseline, 9 months
  One depression scale (range from 0 - 4 with higher values related to worse outcomes)
Change in parent characteristics as assessed by the Parental Modernity Scale | baseline, 9 months
  Two subscales: traditional beliefs (ratings from 1 - 5 with higher values representing traditional beliefs) and progressive beliefs (ratings from 1 - 5 with higher values representing progressive beliefs).
Change in parent characteristics as assessed by the Parenting Stress Index, Fourth Edition Short Form | baseline, 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Janelle J Montroy, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

DOCUMENTS (1):
  • Informed Consent Form (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/45/NCT03431545/ICF_000.pdf